CLINICAL TRIAL: NCT03261154
Title: Serum iPTH, Calcium and Phosphate, and the Risk of Mortality in Beijing Elderly Hemodialysis Population
Status: Completed | Type: Observational
Sponsor: Wenhu Liu (Other)
Responsible Party: Sponsor-Investigator, Wenhu Liu, Director of Nephrology Deptartment, Beijing FH, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: 2016-P2-126-01
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease
Keywords: Serum iPTH; Calcium; Phosphate
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Incidence of End Stage Renal Disease (ESRD) amongst elderly patient group is continuously increasing with population aging progressing. Mineral and bone disorder (MBD) is a common complication caused by ESRD, it raises the incidence of cardiovascular disease (CVD) in hemodialysis patients, as well as mortality.

Joint effects of Kidney failure and aging on elderly hemodialysis patients make the contribution factors of CKD-MBD quite complex, and it also leads to differences in clinic manifestation between elderly hemodialysis patients and non-elderly hemodialysis patients. Since not much studies had been done for this specific subject, thus, research on elderly patients who is taking Maintenance hemodialysis is very necessary. This study is a retrospective research to identify optimized target value of Calcium and Phosphorus for elderly patients taking maintenance hemodialysis and hence provide guidance for clinical practices. The data for this study will be provided by Beijing Blood Purification Quality Control and Improvement Center. Clinical files and Calcium and Phosphorus metabolic indices will be collected amongst elderly patients who were elder than 65 years and was taking maintenance hemodialysis between Jan 1st, 2012 through Dec 31st, 2016. Relationship between Calcium level, Phosphorus level, iPTH index, all-cause mortality and CVD caused mortality will be analyzed to identify optimized range of target Calcium levels, Phosphorus level for hemodialysis treatment

ELIGIBILITY:
Inclusion Criteria:

* The data shall include the information of elderly hemodialysis patients who were 65 years or elder between Jan 1st, 2012 and Dec 31st, 2016

Exclusion Criteria:

* The patients who only has less than 6 months history of hemodialysis since selected in the research patient group The patients who passed away within 3 months since selected in the research patient group The patients who took less than 3 hemodialysis in a week The patients who took kidney transplant during the research time period The patients who do not have blood biochemical results in the records

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: the data for this study will be provided by Beijing Blood Purification Quality Control and Improvement Center. Clinical files and Calcium and Phosphorus metabolic indices will be collected amongst elderly patients who were elder than 65 years and was taking maintenance hemodialysis between Jan 1st, 2012 through Dec 31st, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 5 years
  all patients died in our observation period

SECONDARY OUTCOMES:
CVD-related mortality | 5 years
  the cause of death was cardiovascular disease related

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship hospital, Beijing, Beijing Municipality, China